CLINICAL TRIAL: NCT00211601
Title: Study of Chemotherapy and Patient Health Outcomes for Nausea and Emesis
Brief Title: Study of Chemotherapy and Patient Health Outcomes for Nausea and Emesis (0000-041)
Acronym: C-PHONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0000-041; 041; 2005_072
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting

INTERVENTIONS:
Behavioral: Disease Management Assessment

SUMMARY:
The purpose of this study is to assess whether timely feedback to providers on patient experiences with delayed chemotherapy induced nausea and vomiting (CINV) lead to differences in patient outcomes for subsequent cycles.

ELIGIBILITY:
Inclusion Criteria:

* Highly or moderately emetogenic chemotherapy planned for at least 2 cycles

Exclusion Criteria:

* Concurrent other anti-cancer therapy (e.g. radiation, hormone, etc.); vomiting during the 24 hours prior to first chemotherapy cycle; having a disease/condition or taking medication that may cause emesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2004-08; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
CINV at the delayed phase during cycle 2

SECONDARY OUTCOMES:
Treatment for CINV

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC